CLINICAL TRIAL: NCT04635397
Title: Immunomonitoring After Hematopoietic Stem Cell Transplantation for Hematological Malignancies Using Cytokines Profiling and Flow Cytometry
Brief Title: Immunomonitoring After Hematopoietic Stem Cell Transplantation
Acronym: Allo Monitor
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 20-AOI-05; 2020-A02138-31 (Other: ID RCB)
Record Dates: First submitted 2020-11-06; First posted 2020-11-19 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (HSCT) remains the only curative option for many hematologic malignancies, in particular acute leukemias and myelodysplastic syndromes.

At the center of these reactions are the donor's T and NK cells. Several studies have highlighted the impact of T cells reconstitution on post-transplant infection rates, relapse and GvHD.

Most of the post-allogeneic immune reconstitution studies available to us today include young patients (<60 years of age) who have had genoidentic or phenoidentic 10/10 allografts and mostly only study the phenotype of a limited number of immune cells. While it is important to know the absolute number reconstitution kinetics of the different categories of immune cells, it is essential to also be able to assess the function of the different cells. Knowledge of the restoration of T function at key dates after allogeneic stem cell transplantation would make it possible to adapt post allogeneic immunomodulation (immunosuppressive treatment and injections of donor lymphocytes) and anti-infectious prophylaxis for patients. The measurement of cytokine profiles after nonspecific stimulation of T and NK lymphocytes recently made available to the immunology laboratory of the CHU de Nice allows a routine assessment of T lymphocyte function (Th1, Th2 Th 17 and T regulatory) and NK by measurement of the secretion of different cytokines after stimulation of the patient's lymphocytes with different antigens (anti-CD3 and anti-TLR7).

The cytokine profile during immune reconstitution in hematopoietic cell transplants has never been evaluated; we will analyze it with regard to clinical data: relapse, infections and GVHD.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (HSCT) remains the only curative option for many hematologic malignancies, in particular acute leukemias and myelodysplastic syndromes.

The success of the allogeneic transplant is based on the Graft versus Leukemia (GvL) effect which corresponds to the elimination of tumor cells by the donor's immune system from the recipient's body. Conversely, graft versus host disease (GvHD) is an immune response of the donor versus the host due to major and / or minor histocompatibility differences resulting in multi-organ damage and being the main cause of transplant-related mortality. The main causes of death in allogeneic patients are infections, relapse of the initial disease and GvHD. The relapse linked to an ineffectiveness of the anti-tumor response of the donor's immune system is responsible for 40% of transplant failures. GvHD is present in 40 to 70% of transplants. In both cases, therapeutic options are available in order to modulate the immune response.

In fact, in the event of a relapse of the disease, reinjections of donor lymphocytes make it possible to trigger a GvL effect and cure. For patients with GvHD, on the other hand, treatment is based on increased immunosuppression.

At the center of these reactions are the donor's T and NK cells. Several studies have highlighted the impact of T immune reconstitution on post-transplant infection rates, relapse and GvHD.

Infections and relapses may be linked to insufficient antiviral or anti-tumor responses of the graft (Th1 pathway deficiency) while GvHD is linked to an excessive response of the graft against the host cells (Immune imbalance associating a excess of Th1, Th2 and Th17 responses).

However, there is currently no routine test to predict the kinetics and quality of immune reconstitution in allogeneic patients.

Most of the post-allogeneic immune reconstitution studies available to us today include young patients (<60 years of age) who have had genoidentic or phenoidentic 10/10 allografts and mostly only study the phenotype of a limited number of immune cells. While it is important to know the absolute number reconstitution kinetics of the different categories of immune cells, it is essential to also be able to assess the function of the different cells.

The evaluation of lymphocyte function is mainly based on the measurement of their ability to secrete different cytokines. This measure currently requires complex procedures exclusively reserved for research. Knowledge of the restoration of T function at key dates after allogeneic stem cell transplantation would make it possible to adapt post allogeneic immunomodulation (immunosuppressive treatment and injections of donor lymphocytes) and anti-infectious prophylaxis for patients. The measurement of cytokine profiles after nonspecific stimulation of T and NK lymphocytes recently made available to the immunology laboratory of the CHU de Nice allows a routine assessment of T lymphocyte function (Th1, Th2 Th 17 and T regulatory) and NK by measurement of the secretion of different cytokines after stimulation of the patient's lymphocytes with different antigens (anti-CD3 and anti-TLR7).

The immunology laboratory of the Nice University Hospital recently demonstrated in a cohort of patients with a kidney transplant that the level of secretion of INF-γ (Th1 pathway) by T lymphocytes after non-specific stimulation was correlated with the risk of rejection and inversely correlated with the risk of infectious complications. In addition, in a cohort of patients with an autoimmune disease (Extra-Membranous Glomerulonephritis), the level of secretion of pro-inflammatory cytokines from the Th17 pathway (IL6, IL17, etc.) was correlated with the risk of thrombo-complications. embolic and relapse.

The cytokine profile during immune reconstitution in hematopoietic cell transplants has never been evaluated; we will analyze it with regard to clinical data: relapse, infections and GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Suffering from a malignant hemopathy
* Allogeneic bone marrow or hematopoietic stem cells
* Identical geno-, pheno- and haplo donors
* Informed consent signed by the patient or the person of trust in case of impossibility (deferred consent of the patient when his condition allows it)
* Affiliated with a social security scheme

Exclusion Criteria:

* Patient with a clinical or biological contraindication to performing an allogeneic transplant
* Patient with progressive solid cancer or in remission for less than 3 years
* HIV-positive patients
* Patients with chronic active hepatitis B or C
* Allogeneic cord blood transplant
* Allograft with sequential conditioning
* Post-allograft preemptive treatment other than injections of donor lymphocytes Withdrawal of informed consent
* Inability to undergo medical monitoring of the study for geographical, social or psychological reasons

Non-inclusion criteria:

* Minor patient
* Pregnant woman
* Patient with congenital or previously acquired immune deficiency
* Patient on prior immunosuppressive treatment
* Patient under guardianship or guardianship or placed in detention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving an allogeneic stem cell transplantation for an hematological malignancy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-02-03 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2026-08-18 (Estimated)

PRIMARY OUTCOMES:
Qualitative and quantitative evaluation of T and NK lymphocyte reconstitution in post allogeneic transplant | on day 2 post transplant,
  measuring cytokine profiles (Th1, Th2 or Th17) after non-specific stimulation of T and NK lymphocytes
Qualitative and quantitative evaluation of T and NK lymphocyte reconstitution in post allogeneic transplant | 90 days post transplant,
  measuring cytokine profiles (Th1, Th2 or Th17) after non-specific stimulation of T and NK lymphocytes
Qualitative and quantitative evaluation of T and NK lymphocyte reconstitution in post allogeneic transplant by measuring cytokine profiles (Th1, Th2 or Th17) after non-specific stimulation of T and NK lymphocytes | 6 months
  measuring cytokine profiles (Th1, Th2 or Th17) after non-specific stimulation of T and NK lymphocytes
Qualitative and quantitative evaluation of T and NK lymphocyte reconstitution in post allogeneic transplant | one year after allogeneic transplantation
  measuring cytokine profiles (Th1, Th2 or Th17) after non-specific stimulation of T and NK lymphocytes
Qualitative and quantitative evaluation of T and NK lymphocyte reconstitution in post allogeneic transplant | in the event of a proven relapse or occurrence of acute grade 2 or more GVHD
  measuring cytokine profiles (Th1, Th2 or Th17) after non-specific stimulation of T and NK lymphocytes

SECONDARY OUTCOMES:
Overal | at Day 90 post allograft
relapse-free survival | at Day 90 post allograft
Overall | Month 6 post allograft,
relapse-free survival | Month 6 post allograft,
Overall | Month 12 post allograft
relapse-free survival | Month 12 post allograft
Incidence of acute GvH | Day 90 post allograft
Incidence of acute GvH | Month 6 post allograft
Incidence of chronic GvH | at Day 90, Month 6 and Month 12 post transplant
Incidence of relapses | at Day 90, Month 6 and Month12 post transplant
Incidence of infectious events | Day 90, Month 6 and Month 12 post transplant
Quantification of T, B and NK lymphocyte populations by flow cytometry already performed as part of the management of allogeneic patients | during the study
Study the correlation between the measurement of cytokine profiles (Th1, Th2 or Th17) after nonspecific stimulation of T and NK lymphocytes | on day 2 post transplant, 90 days post transplant, 6 months and one year post allogeneic transplant and in the event of proven relapse. or occurrence of acute grade 2 or greater GVHD and other secondary endpoints

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, CHU de NICE, France

IPD SHARING:
Plan to Share IPD: No